CLINICAL TRIAL: NCT00038558
Title: Prophylactic Use of Filgrastim SD/01 In Patients With Hodgkin's Disease Receiving ABVD Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID01-087
Record Dates: First submitted 2002-05-31; First posted 2002-06-03 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Hodgkin Disease
Keywords: Hodgkin's lymphoma; Dacarbazine; DTIC; DTIC-Dome; Vinblastine; Velban; Bleomycin sulfate; Blenoxane; BLM; Doxorubicin Hydrochloride; Adriamycin; Filgrastim; G-CSF; Neupogen; Pegfilgrastim; granulocyte colony-stimulating factor
MeSH Terms: conditions — Hodgkin Disease | interventions — pegfilgrastim; Granulocyte Colony-Stimulating Factor; Filgrastim; Doxorubicin; Bleomycin; Vinblastine; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Filgrastim + ABVD Chemotherapy (Experimental)
  Interventions: Drug: Filgrastim SD/01; Drug: Adriamycin; Drug: Bleomycin; Drug: Vinblastine; Drug: DTIC

INTERVENTIONS:
Drug: Filgrastim SD/01
  Other Names: G-CSF; Neupogen
Drug: Adriamycin
  Other Names: Doxorubicin Hydrochloride; Adriamycin PFS; Adriamycin RDF
Drug: Bleomycin
  Other Names: Bleomycin sulfate; Blenoxane; BLM
Drug: Vinblastine
  Other Names: Velban
Drug: DTIC
  Other Names: DTIC-Dome; Dacarbazine

SUMMARY:
Prophylactic use of Filgrastim SD/01 for patients with Hodgkin's lymphoma receiving ABVD chemotherapy.

ELIGIBILITY:
INCLUSION:

* Previously untreated Hodgkin's disease patients who are scheduled to receive standard ABVD chemo.
* Histologically proven diagnosis of Hodgkin's disease of any type.
* Bidimensionally measurable disease.
* Signed informed consent.
* Age >/= 16 yrs.
* Adequate bone marrow reserve (ANC>1000/uL, Platelet >100,000/uL.
* LVEF>/=50% by MUGA scan or echocardiogram.
* Serum creatinine <2mg/dL; serum bilirubin<2mg/dL.

EXCLUSION:

* HIV positive.
* Pregnant women and those of child bearing age who are not using adequate contraception.
* Prior chemotherapy.
* Severe pulmonary disease including COPD and asthma.
* History of prior sensitivity to E.coli derived products.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2001-11; Primary Completion 2004-02 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Response to Prophylactic Filgrastim SD/01Chemotherapy | Following ABVD chemotherapy course

CONTACTS AND LOCATIONS:
Overall Officials: Anas Younes, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org